CLINICAL TRIAL: NCT00668889
Title: Dermatological Evaluation of the Photo Irritation and Photo Sensitivity Potential for Dermacyd Tina Gel Tangerina Mix.
Brief Title: Dermacyd Tina Gel Tangerina Mix - Photo Evaluation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: GMA-CO/Medical Director, sanofi-aventis administrative office France
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACAC_L_03737
Record Dates: First submitted 2008-04-23; First posted 2008-04-29 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: Hygiene
MeSH Terms: interventions — Lactic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lactic acid (Dermacid)

SUMMARY:
The purpose of this study is to prove the absence of photo irritation and photo sensitivity potential of the product Dermacyd Tina Gel Tangerina Mix.

ELIGIBILITY:
Inclusion Criteria:

* Phototype Skin II and III
* Integral skin test in the region

Exclusion Criteria:

* Lactation or gestation
* Use of Antiinflammatory and/or immunosuppression drugs 15 days before the selection
* Diseases which can cause immunity decrease, such as HIV, diabetes
* Use of drug photosensitizer
* History of sensitivity or irritation for topic products
* Active cutaneous disease which can change the study results
* History or photodermatosis active
* Family or personal antecedent of cutaneous photoinduced neoplasias
* Presence of a precursor lesion of cutaneous neoplasia, such as nevus melanocyte and keratoses actinium
* Intense solar exposure in the study area
* Use of new drugs or cosmetics during the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The photo irritation test and the photosensitivity will be measured using UVA irradiation and evaluated according International Contact Dermatitis Research Group (ICDRG) scale. The sensibility will be evaluated according to the skin type. | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi-aventis administrative office Brazil
Locations (1):
- Sanofi-aventis administrative office, São Paulo, São Paulo, Brazil